CLINICAL TRIAL: NCT03127891
Title: Effect of Short Term Pranayama on Anaesthesia Management in Patients Undergoing Cardiac Surgery
Brief Title: Effect of Yoga on Anesthesia Management
Acronym: yoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, aspari mahammad azeez, Junior resident, dept.of anesthesia and intensive care, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NK/3047/MD/807
Record Dates: First submitted 2017-01-08; First posted 2017-04-25 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Anesthesia; Closed Loop Anesthesia Delivery System (CLADS)
Keywords: pranayama yoga
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pranayama yoga (Experimental): yoga breathing exercise
  Interventions: Behavioral: pranayama yoga
- control group (Placebo Comparator): no intervention
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: pranayama yoga — providing short term pranayama yoga for 5 sessions before surgery patients under going cardiac surgery.
  Other Names: yoga breathing exerxises
  Arms: pranayama yoga
Other: control group — no intervention should be given to patients allocated to this group
  Arms: control group

SUMMARY:
TITLE: EFFECT OF SHORT-TERM PRANAYAMA ON ANAESTHESIA MANAGEMENT IN PATIENTS UNDERGOING CARDIAC SURGERY

Primary aim: To evaluate the effect of pre-operative short term pranayama yoga on stress-induced hemodynamic (HR, MAP) changes in patients scheduled for cardiac surgery.

Secondary aims:

1. To compare the effect of YOGA on preoperative anxiety.
2. To compare the effect of Yoga on SPO2.
3. To compare effect of Yoga on total consumption of propofol administered using Closed Loop Anaesthesia Delivery system(CLADS)
4. To compare effect of Yoga on total consumption of fentanyl, and vecuronium
5. To compare effect of Yoga on post-operative anxiety (after extubation in CTVS ward)
6. To compare effect of Yoga on postoperative outcome in terms of duration of mechanical ventilation, duration of ICU stay, incidence of complications and post-op mortality

DETAILED DESCRIPTION:
TITLE: EFFECT OF SHORT-TERM PRANAYAMA ON ANESTHESIA MANAGEMENT IN PATIENTS UNDERGOING CARDIAC SURGERY

This will be a prospective randomized controlled pilot study. After Institutional Ethics Committee approval and written informed consent patients aged 20-60 years and scheduled for elective cardiac surgery will be assessed for eligibility.

All patients admitted in the CT VS ward and awaiting elective surgery in the next 5-6 days will be recruited. The patients will be divided randomly into two groups using random number table; Group C: Control, Group Y: Yoga. Allocation will be done using sealed envelope technique. The study will be conducted from October 2016 to December 2017.

Before any intervention the baseline haemodynamic parameters will be recorded and general anxiety score will be measured using Spielberg's state-trait anxiety inventory (STAI).

Group Y:

Yoga sessions will be held for the patients during their hospitalization in the CTVS ward in the evening in a dedicated YOGA room. A YOGA instructor will train the patients for the YOGA sessions. Target is to give a minimum of 5 sessions of YOGA in this group of patient. yoga training will be done for 60 min. The vital signs (HR, BP, and SPO2)of the patients before and after each session will be recorded using multi-parameter vital sign monitors.

Anulom Vilom Pranayam: (10 min)

The patient will be asked to sit comfortably and close his eyes.

* Close the right nostril with the right thumb
* Inhale slowly through the left nostril and fill lungs with air.
* Close left nostril with the ring and middle fingers of the right hand and open the right nostril.
* Exhale slowly and completely with the right nostril.
* Again inhale through the right nostril and fill lungs.
* Close the right nostril by pressing it with the right thumb.
* Open the left nostril, breathe out slowly. Udgith Pranayama (10 min )

  1. The patient will be made to sit in a comfortable posture with spine erect and in line with neck and head.
  2. He/She will be instructed to put the hands in Gyan mudra and eyes closed.
  3. Being aware of their breath, the participant will be instructed to breathe deeply through the nose.
  4. During exhalation "AUM" will be chanted for as long as their body allows.The participant will not be stressed.

Nadishodhana Pranayama (10 minutes)

1. The patient will be made to sit in a comfortable posture with spine erect and in line with neck and head
2. The participant will be instructed to fold the index finger and middle finger of the right hand in such a way that their tips touch the root of the right thumb. The ring finger and little finger of right hand will be extended and placed on the left nostril. Right thumb will be placed on right nostril
3. The participant will be made to close the eyes.
4. The right nostril will be closed and deep inhalation will be taken from the left nostril.
5. The left nostril will be closed and exhalation will be carried out through the right nostril.
6. Inhalation will be done through right nostril keeping the left nostril closed.
7. Exhalation will be done through left nostril keeping the right nostril closed.
8. This will complete one round.

Sheetali (5 min) The patients will be made to sit in a comfortable posture with spine erect and in line with neck and head.Eyes will be closed gently.

1. The patients will be instructed to open their mouth and stretch the tongue as long as he/she can.
2. The tongue will be rolled from sides such that tongue takes the form of a hollow tube.
3. Air will be inhaled through this hollow tube.
4. Later, the mouth will be closed and exhalation will be carried out through the nose.

Bhramari Pranayama ( 10 min )

1. The patients will be made to sit in a comfortable posture with spine erect and in line with neck and head.Eyes will be closed gently.
2. The hands will be preferably kept in Shanmukhi mudra. If not comfortable, Gyan mudra will have opted and eyes will be kept closed.
3. Being aware of their breath, the participant will be instructed to breathe deeply through nose
4. During exhalation, humming sound will be produced for as long as the participant's body allows. They will not be stressed.
5. The vibration generated within the body will be felt.

YogNidra / Relaxation (15 min)

The participant will be made to lie down in Shavasana and made to follow the instructions.

Group C;

Patients in this group will not be given any yoga session and will thus act as a control group. The vital signs (HR, BP, and SPO2)of the patients will be recorded using multi-parameter vital sign monitors for the subsequent days after recruitment and group allocation.

Anesthetic management for cardiac surgery:

Anxiety score will be measured by using the State-Trait Anxiety Inventory (STAI) on the day of surgery. The hemodynamic parameters will be recorded for subsequent comparison of the effect of Yoga.

This will be followed by insertion of a 16 G i.v cannula after giving local anesthetic with a 26 G needle. Following monitors will be attached: continuous pulse oximetry (SpO2), electrocardiogram (ECG), periodic non-invasive blood pressure (S/Anesthesia monitor, Datex Ohmeda Inc., Madison, WI), and continuous BIS (BIS XP, Aspect Medical Systems, Newton, MA in the S/5 Anesthesia monitor). Pre-induction arterial line and the central line will be secured in all patients after giving local anesthetic and continuous arterial blood pressure and central venous pressure measurements will be recorded.

Induction of anesthesia will be performed with propofol using closed-loop anesthesia delivery system (CLADS) titrated to target BIS of 50 and fentanyl 3 mcg/kg in both groups. Muscular paralysis for tracheal intubation will be achieved by vecuronium bromide 0.1mg/kg followed by intermittent boluses. After intubation, volume-controlled mechanical ventilation to be provided with FiO2 0.5, tidal volume 7-8 ml/kg, positive end-expiratory pressure (PEEP) 5 cm H2O, and respiratory rate of 12-14/min. Patients will be mechanically ventilated with air: oxygen mixture (50:50) to maintain end-tidal carbon dioxide (ETCO2) values between 30 and 35 mm Hg. Maintenance of anesthesia will be done with propofol infusion using CLADS titrated to target BIS value of 40-60. Fentanyl infusion at 1.0 mcg/kg/h will be administered for analgesia. Fentanyl 1 mcg/kg will be administered before sternotomy. Nasopharyngeal temperature, urinary output, and ETCO2 will be recorded. CPB will be initiated after heparinization with an intravenous dose of 3 mg/kg titrated to the ACT of 450 seconds.Every 20 min, cardioplegia will be repeated. The MAP will be maintained in the range 50-70 mm Hg during CPB. Weaning from CPB will be performed in a stepwise manner. Appropriate inotropes adrenaline/ noradrenaline/ dopamine/ milrinone will be used to maintain adequate tissue perfusion and cardiac output. Fluid replacement will include crystalloid solutions with an initial infusion rate 6-7 ml.kg.hr prior to and during anesthesia and 2- 3 ml/kg/hr postoperatively. All the anesthesia drug consumption data will be recorded online using CLADS.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-60y
* Cardiac surgery( valvular heart disease and coronary artery disease)

Exclusion Criteria:

* Severe restrictive lung disease
* Severe obstructive lung disease
* NYHA-4
* Drug addicts
* History of smoking
* Alcohol intake
* Central nervous system disease
* Psychiatric disorder

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11; Primary Completion 2018-05-20 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
The effect of pre-operative short term pranayama yoga on heart rate in patients scheduled for cardiac surgery. Measuring heart rate by using clarity ARGUS LCM PLUS multi - parameter monitor. | minimum 5 days
  Heart rate will be measured before and after every yoga session for 5 consecutive days
The effect of pre-operative short term pranayama yoga on mean arterial pressure in patients scheduled for cardiac surgery. Measuring mean arterial pressure using clarity ARGUS LCM PLUS multi - parameter monitor. | Minimum 5 days
  Mean arterial pressure will be measured before and after every yoga session for 5 consecutive days
The effect of pre-operative short term pranayama yoga on SpO2 in patients scheduled for cardiac surgery. Measuring SpO2 using clarity ARGUS LCM PLUS multi - parameter monitor. | Minimum 5 days
  SpO2 will be measured before and after every yoga session for 5 consecutive days

SECONDARY OUTCOMES:
the effect of YOGA on pre operative anxiety. pre operative anxiety will be measured by STAI (state and trait anxiety inventory) scale | minimum 5 days preoperatively
  pre operative anxiety will be measured by STAI scale before first yoga session and after last yoga session
consumption of propofol | approx 8-12hrs
  intra operative consumption of opioid propofol consumption during induction and maintenance of anesthesia
Fentanyl consumption | approx 8-12 hrs
  intra operative consumption of opioid fentanyl consumption during induction and maintenance of anesthesia
vecuronium consumption | approx 8-12 hrs
  intra operative consumption of muscle relaxant vecuronium during induction and maintenance of anesthesia
post-operative anxiety. Post operative anxiety will be measured by STAI (state and trait anxiety inventory) scale | at 12 hrs after extubation
  will be measured by using STAI score 12 hours after extubation
post-operative outcome (complications) | approx 7 days
  post operative complications related to surgery and anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Goverdhan D Puri, MD,PhD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Aspari Mahammad Azeez, Chandigarh, Apmc 77179, India

IPD SHARING:
Plan to Share IPD: No